CLINICAL TRIAL: NCT00030381
Title: Phase I Trial of 4'-IODO-4'-Deoxydoxorubicin in Primary Amyloidosis (AL)
Brief Title: Iododoxorubicin in Treating Patients With Primary Systemic Amyloidosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02443; MC0113; U01CA069912 (NIH); CDR0000069160 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-02-14; First posted 2003-09-17 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Primary Systemic Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — 4'-deoxy-4'-iododoxorubicin

ARMS (1):
- Treatment (iododoxorubicin) (Experimental): Patients receive iododoxorubicin IV over 15 minutes on days 1, 8, 15, and 22. Treatment repeats every 12 weeks for a total of 4 courses or a cumulative dose of 400 mg/m^2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 4'-iodo-4'-deoxydoxorubicin; Other: pharmacological study

INTERVENTIONS:
Drug: 4'-iodo-4'-deoxydoxorubicin — Given IV
  Other Names: IDOX; iododoxorubicin
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Iododoxorubicin may dissolve protein deposits and be an effective treatment for primary systemic amyloidosis. Phase I trial to determine the effectiveness of iododoxorubicin in treating patients who have primary systemic amyloidosis

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of iododoxorubicin in patients with primary systemic amyloidosis.

SECONDARY OBJECTIVES:

I. Determine the safety, especially cardiac safety, of this drug in these patients.

II. Determine the survival rate of patients treated with this drug. III. Determine, preliminarily, the clinical efficacy of this drug in these patients.

IV. Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive iododoxorubicin IV over 15 minutes on days 1, 8, 15, and 22. Treatment repeats every 12 weeks for a total of 4 courses or a cumulative dose of 400 mg/m^2 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of iododoxorubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histochemically confirmed amyloidosis by polarizing microscopy of greenbirefringent material in Congo red-stained tissue specimens
* At least one of the following:

  * Demonstrable M-protein in serum or urine
  * Clonal population of plasma cells in bone marrow
  * Immunohistochemical stain with anti-light chain antisera of amyloid fibrils
* Symptomatic organ involvement, including liver involvement, mild cardiac involvement, renal involvement, grade 1 or 2 peripheral neuropathy, or soft tissue involvement (including tongue)

  * No purpura or carpal tunnel syndrome as sole manifestation of disease
* No clinically overt multiple myeloma defined as monoclonal bone marrow platelet concentration greater than 20% and at least one of the following:

  * Bone lesions
  * Anemia
  * Hypercalcemia
* Performance status - ECOG 0-3 (3 allowed only if related to muscular infiltration by amyloid or peripheral neuropathy)
* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Total bilirubin no greater than 2.0 mg/dL
* Direct bilirubin no greater than 1.0 mg/dL
* Alkaline phosphatase no greater than 4 times upper limit of normal (ULN)
* AST or ALT no greater than 3 times ULN
* Creatinine clearance at least 40 mL/min
* Ejection fraction at least 50% by echocardiogram
* No New York Heart Association class III or IV heart disease
* No enzyme-documented myocardial infarction within the past 3 years
* No chronic atrial fibrillation
* No grade 2 or 3 atrioventricular block (Mobitz type I allowed)
* No sustained (greater than 30 seconds) ventricular tachycardia, more than 1 episode of non-sustained ventricular tachycardia (3 consecutive ventricular beats), or frequent (more than 20 in 24 hours) ventricular pairs by 24-hour ambulatory electrocardiographic monitoring
* No intraventricular septum greater than 16 mm by echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No other active malignancy except nonmelanoma skin cancer or cervical cancer
* No psychiatric illness or social situation that would preclude study
* No severe diarrhea (greater than grade 3) that is not controllable with medication or that requires total parenteral nutrition
* More than 4 weeks since prior interferon alfa
* No concurrent immunotherapy
* More than 4 weeks since prior melphalan or other alkylating agents
* No prior anthracycline exposure greater than 120 mg/m^2
* Recovered from prior chemotherapy
* No other concurrent chemotherapy
* More than 4 weeks since prior high-dose dexamethasone
* No concurrent radiotherapy
* No concurrent investigational ancillary therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-12; Primary Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
MTD of IDOX defined as the highest safely-tolerated dose where =< 1 patient experiences DLT with the next higher dose having at least 2 patients who experience DLT | 12 weeks
  The number and severity of toxicity incidents will indicate the level of tolerance of IDOX in the treatment of primary amyloidosis. Non-hematologic toxicities will be evaluated via the ordinal CTC standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir and percent change from baseline values) as well as categorization via CTC standard toxicity grading.

SECONDARY OUTCOMES:
Laboratory correlates | Up to 3 months post treatment
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures will be carried out by standard parametric and non-parametric correlation procedures (Pearson's and Spearman's coefficients). Prerequisite normality testing of these data will be carried out via standard Shapiro and Wilk (25) testing.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States